CLINICAL TRIAL: NCT06762379
Title: Implementation of a New Algorithm for HRR Gene Mutation Testing in Patients With mPC
Brief Title: Implementation of a New Algorithm for HRR Gene Mutation Testing in Patients With mPC Through Liquid Biopsy Integration
Acronym: L2-267
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: L2-267
Record Dates: First submitted 2024-12-31; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Metastatic Prostate Cancer (mPC)
Keywords: HRR liquid biopsy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Biospecimen Retention: Samples With DNA — blood, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient with metastatic prostate cancer (mPC)

SUMMARY:
Implementation of a new algorithm for HRR gene mutation testing in patients with mPC through liquid biopsy integration

DETAILED DESCRIPTION:
Analysis of the current clinical landscape of mPC Italy to identify gaps and opportunities for improvement.

Patient identification and enrollment Blood sample collection and plasma purification ctDNA extraction and NGS analysis of homologous recombination repair (HRR) genes. Clinical Real-World Data (RWD) and molecular analysis data collection Testing algorithm development based on collected data Finalization and sharing of a best practice model for diagnostic procedures in mPC patients

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic prostate cancer whose tumor tissue is unavailable or inadequate for molecular testing. • Written informed consent must be signed and dated by the patient and the investigator prior to inclusion.

Exclusion Criteria:

* Unable to provide written informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Validation of an assay for homologous recombination repair (HRR) gene mutation testing using liquid biopsy | 3 years
  Validation of an assay for homologous recombination repair (HRR) gene mutation testing using liquid biopsy in patients with metastatic prostate cancer (mPC) whose tumor tissue is inadequate or unavailable for molecular testing.

CONTACTS AND LOCATIONS:
Locations (1):
- European Institute of oncology, Milan, Italy